CLINICAL TRIAL: NCT01024387
Title: A Multi-Institutional, Phase II Open-Label Study of AMG 479 in Advanced Carcinoid and Pancreatic Neuroendocrine Tumors
Brief Title: AMG 479 in Advanced Carcinoid and Pancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Amgen (Industry)
Responsible Party: Principal Investigator, Matthew H. Kulke, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-240
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Neuroendocrine Tumor; Carcinoid Tumor; Pancreatic Neuroendocrine Tumor
Keywords: AMG 479
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell | interventions — ganitumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMG 479 (Experimental): Patients receive AMG 479 at a dose of 18 mg/kg administered IV on day 1 (± 3 days) of every 3-week cycle. Treatment should continue until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: AMG 479

INTERVENTIONS:
Drug: AMG 479
  Other Names: ganitumab

SUMMARY:
The purpose of this research study is to determine the effectiveness of AMG 479 against carcinoid and pancreatic neuroendocrine tumors. AMG 479 is an antibody that is made in the laboratory. Antibodies are highly specific proteins produced by the body's immune system that recognize foreign substances in the body. AMG 479 has been used in other research studies and information from those other research studies suggests that AMG 479 may help to prevent the growth of some neuroendocrine tumors. The observed antitumor activity of AMG 479, together with the current limited treatment options available for patients with neuroendocrine tumors, warrant further investigation of AMG 479 in this patient population.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) comprise a heterogeneous spectrum of neoplasms. NETs are commonly subclassified into two broad subgroups according to their site of origin: pancreatic NETs are thought to arise from the endocrine cells of the pancreas, whereas NETs of other sites such as the lungs or gastrointestinal tract are often referred to as carcinoid tumors. While histologically similar, carcinoid tumors and pancreatic neuroendocrine tumors have demonstrated different response rates in prior phase II studies of antitumor agents. Because of these differences, we will perform the current study using two cohorts of patients (30 with carcinoid and 30 with pancreatic neuroendocrine tumors). The statistical design, however, is the same for both cohorts. With 30 patients in each cohort, this study has 80% power assuming type I error of 6% to differentiate a >/=17% objective response rate from a </=5% objective response rate using a single stage design. The proposed regimen would be promising in either cohort if at least 4 of 30 patients achieve an objective response.

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic carcinoid or pancreatic neuroendocrine tumors. To be classified as having a pancreatic neuroendocrine tumor, patients must have clinical evidence of currently having or having had a primary pancreatic neuroendocrine lesion.
* Measurable disease by RECIST criteria
* Evidence of progressive disease (by RECIST) within 12 months of study entry.
* Tumors must be considered well- or moderately-differentiated. Patients with poorly differentiated neuroendocrine carcinoma of small cell carcinoma are excluded from this study.
* Adequate hepatic, renal, bone marrow and glycemic function as outlined in the protocol
* Prior treatment with chemotherapy, hepatic artery embolization, surgery or other therapeutic agents is allowed.
* Prior or concurrent therapy with somatostatin analogs is permitted: however patients must continue on a stable dose of somatostatin analogs while receiving study treatment.
* 18 years of age or older
* ECOG performance status 0, 1, or 2 [Eastern Cooperative Oncology Group ]
* Life expectancy of at least 12 weeks
* Negative pregnancy test
* Ability to sign informed consent

Exclusion Criteria:

* Poorly differentiated or small cell neuroendocrine carcinomas
* Insulin secreting pancreatic neuroendocrine tumors (insulinomas)
* Clinically apparent central nervous system metastases or carcinomatous meningitis.
* Myocardial infraction in the past 6 months
* Major surgery 4 weeks prior to enrollment
* Uncontrolled serious medical or psychiatric illness
* Pregnant or lactating women. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study.
* Prior antitumor therapy within 4 weeks of enrollment (with the exception of somatostatin analogs).
* Recent infection requiring systemic anti-infective treatment that was completed 14 days or less prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection).
* Known positive test for human immunodeficiency virus, hepatitis C, chronic or active hepatitis B
* Prior IGF or IGF receptor inhibitor therapy [insulin like growth factor ]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Strosberg JR, Chan JA, Ryan DP, Meyerhardt JA, Fuchs CS, Abrams T, Regan E, Brady R, Weber J, Campos T, Kvols LK, Kulke MH. A multi-institutional, phase II open-label study of ganitumab (AMG 479) in advanced carcinoid and pancreatic neuroendocrine tumors. Endocr Relat Cancer. 2013 May 21;20(3):383-90. doi: 10.1530/ERC-12-0390. Print 2013 Jun. PMID 23572164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from June 2010 through June 2011.
Period: Overall Study
Arm/Group | AMG 479
Started | 60
Evaluable for PFS (One of the patients uneval for resp was incl in PFS eval dataset which included follow-up for death.) | 54
Evaluable for Response (symptomatic deterioration (n=2), patient or MD decision (n=2 each), hypersensitivity reaction (n=1)) | 53
Completed (Given treatment duration is not fixed, all patients are considered as 'Non Completed'.) | 0
Not Completed | 60
Not completed — Radiographic Progression | 29
Not completed — Symptomatic Progression | 10
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 5
Not completed — Death | 2
Not completed — Prolonged Treatment Delay | 1
Not completed — Adverse Event | 3
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Arm/Group | AMG 479
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate is the percentage of patients achieving partial response (PR) or complete response (CR) per RECIST 1.0 criteria. For target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR or PR status must be confirmed by repeat assessments performed no fewer than 4 weeks or more than 6 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline, every 3 cycles (9 weeks) on treatment and at end of treatment. Patients in this study cohort received a median of 6 treatment cycles (18 weeks).
Population: The analysis dataset is comprised of all response evaluable patients.
Measure: Number; unit: percentage of patients
Arm/Group | AMG 479
Number analyzed (Participants) | 53
percentage of patients | 0.0

2. Secondary Outcome: Duration of Response
Description: The duration of response is measured from the time measurement criteria are met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: as for outcome 1
Population: This endpoint was not evaluated because zero patients achieved objected response per RECIST criteria.
Arm/Group | AMG 479
Number analyzed (Participants) | 0

3. Secondary Outcome: Grade 3-4 Toxicity Rate
Description: Grade 3-4 toxicity rate is the percentage of patients who experienced a grade 3 or 4 adverse event with treatment attribution of possible, probable or definite based on CTCAEv4.
Time Frame: Toxicity was evaluated every cycle (3 weeks) on treatment. Patients in this study cohort received a median of 6 treatment cycles (18 weeks).
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | AMG 479
Number analyzed (Participants) | 60
percentage of patients | 31.7 [22.3 to 45.0]

4. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) based on the Kaplan-Meier method is defined as the time from the start of treatment to the date of the first documented disease progression or death due to any cause. Patients without an event were censored at the earliest date of last disease assessment or initiation of non-protocol anti-cancer therapy. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline, every 3 cycles (9 weeks) on treatment and at end of treatment. Patients in this study cohort were followed up to 20 months.
Population: The analysis dataset is comprised of all PFS evaluable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 479
Number analyzed (Participants) | 54
months | 6.3 [4.2 to 12.6]

5. Secondary Outcome: 1-Year Overall Survival
Description: Overall survival (OS) based on the Kaplan-Meier method is defined as the time from treatment start to the date of death or censored at the date last known alive. 1-year overall survival is the probability (%) of remaining alive 1 year from the start of treatment.
Time Frame: Patients in this study cohort were followed up to 20 months.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | AMG 479
Number analyzed (Participants) | 60
percent probability | 66 [52 to 77]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were evaluated every cycle (3 weeks) on treatment. Patients in this study cohort received a median of 6 treatment cycles (18 weeks).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Arm/Group | AMG 479
Serious Adverse Events (participants affected / at risk) | 19/60
Other Adverse Events (participants affected / at risk) | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 479 (N=60)
Anemia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Infusion related reaction (General disorders) | 1
Lung infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Alkaline phosphatase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 479 (N=60)
Anemia (Blood and lymphatic system disorders) | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Spleen disorder (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 4
Hearing impaired (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Cushingoid (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 22
Anal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 3
Cecal hemorrhage (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 4
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 6
Gastric fistula (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 3
Malabsorption (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 21
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal fistula (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Rectal pain (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Chills (General disorders) | 10
Death NOS (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 34
Fever (General disorders) | 9
Flu like symptoms (General disorders) | 1
Hypothermia (General disorders) | 1
Infusion related reaction (General disorders) | 8
Irritability (General disorders) | 1
Malaise (General disorders) | 6
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 5
Sudden death NOS (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 7
Allergic reaction (Immune system disorders) | 3
Abdominal infection (Infections and infestations) | 1
Anorectal infection (Infections and infestations) | 2
Bronchial infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Infections and infestations - Other, specify (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 2
Burn (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 6
Creatinine increased (Investigations) | 3
INR increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 15
Weight loss (Investigations) | 10
White blood cell decreased (Investigations) | 6
Investigations - Other, specify (Investigations) | 1
Alcohol intolerance (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 10
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 24
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypoglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 7
Confusion (Psychiatric disorders) | 3
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 11
Psychiatric disorders - Other, specify (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 2
Uterine pain (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2
Flushing (Vascular disorders) | 5
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 5
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No